CLINICAL TRIAL: NCT07296263
Title: Evaluation of Gadolinium Based Contrast Agents for Portable MR Imaging Systems
Acronym: Contrast PMR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hyperfine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20254565
Record Dates: First submitted 2025-12-17; First posted 2025-12-22 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Intra-axial Tumors; Extra-axial Tumors; Infection/Inflammatory Lesions
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: The Swoop® Portable MR Imaging® System was originally cleared by the U.S. Food and Drug Administration (FDA) on February 6, 2020, under 510(k) number K192002, and has undergone several FDA-cleared updates since its initial clearance. The most recent update was cleared on May 30, 2025, under 510(k) number K250236. All hardware used in this study will be covered under one of these FDA clearances. However, certain imaging sequences utilized for research purposes may be investigational and are not part of the cleared indications for use. The intent of the study is to demonstrate the established benefits of gadolinium-based contrast agents are observable in T1W images at 64 mT. All systems used will be FDA cleared hardware. Investigational-use only imaging sequences may be used for image collection; however, all hardware-imposed safety limitations will remain in place.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Evaluation of Gadolinium Based Contrast Agents for Portable MR Imaging Systems (Other): This prospective, interventional, single-arm study will collect data from patients in the hospital and/or outpatient setting undergoing portable magnetic resonance imaging (pMRI) using the Swoop® Portable MR Imaging® System (0.064 T). Each participant will undergo a pre-contrast portable MRI (pMRI) imaging scan, followed by intravenous administration of an FDA approved gadolinium-based contrast agent (GBCA), and then complete a post-contrast pMRI imaging scan. The study will assess lesion visibility between pre- and postcontrast images to assess the added value of contrast enhancement.
  Interventions: Other: Evaluation of Gadolinium Based Contrast Agents (GBCA) for Portable MR Imaging Systems

INTERVENTIONS:
Other: Evaluation of Gadolinium Based Contrast Agents (GBCA) for Portable MR Imaging Systems — This prospective, interventional, single-arm study will collect data from patients in the hospital and/or outpatient setting undergoing portable magnetic resonance imaging (pMRI) using the Swoop® Portable MR Imaging® System (0.064 T). Each participant will undergo a pre-contrast portable MRI (pMRI) imaging scan, followed by intravenous administration of an FDA approved gadolinium-based contrast agent (GBCA), and then complete a post-contrast pMRI imaging scan. The study will assess lesion visibility between pre- and postcontrast images to assess the added value of contrast enhancement.

SUMMARY:
This is a prospective, multi-center, interventional study designed to evaluate the visualization benefits of FDA approved gadolinium-based contrast agents (GBCAs) in portable magnetic resonance imaging (pMRI) of the brain. The study will enroll adult patients with known or suspected brain lesions involving blood-brain barrier disruption. Each participant will undergo a pre-contrast pMRI scan, receive an intravenous GBCA injection, and then complete a post-contrast pMRI scan using the Swoop® Portable MR Imaging® System. Lesion visualization will be assessed by independent neuroradiologists using standardized scoring criteria. The study will be conducted across a minimum of three sites to ensure diversity in patient population, imaging environments, and GBCA types.

ELIGIBILITY:
Inclusion Criteria:

* Study inclusion criteria:

Subjects must meet ALL of the following inclusion criteria to be eligible for enrollment:

1. Age ≥18 years.
2. Clinical target: Highly suspected brain lesion(s) with focal blood-brain barrier disruption (preferably documented on prior standard-of-care high-field MRI within the past 60 days).
3. MRI/contrast approval: Cleared for pMRI and for approved IV GBCA administration per site policy.
4. IV access: Adequate peripheral venous access for contrast injection.
5. Consent/participation: Able to provide informed consent and comply with brief supine imaging (pre- and postcontrast).

Exclusion Criteria:

* Subjects must not meet ANY of the following Exclusion criteria to be eligible for enrollment:

  * Metallic clips or devices in the brain or eye.
  * Body weight greater than 200 kg. Inability to fit or be positioned appropriately within the Swoop® Portable MR Imaging® System.
  * Inability to remain still or lie flat during the imaging period.
  * Not cleared for GBCA administration due to known hypersensitivity, allergy, or contraindication.
  * Severe renal impairment (eGFR < 30 mL/min/1.73 m²) or acute kidney injury.
  * History of severe reaction to any gadolinium-based contrast agent.
  * Known or suspected pregnancy at the time of imaging.
  * Any medical or behavioral condition that, in the investigator's judgment, would make participation unsafe or interfere with study completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Radiologist-rated lesion border delineation on post-contrast portable MRI | 6 months
  Blinded neuroradiologists will assess lesion border delineation on post-contrast T1-weighted portable MRI images using a standardized 5-point Likert scale (1 = poor delineation, 5 = excellent delineation). Scores will be summarized using descriptive statistics.
Radiologist-rated lesion internal morphology visibility on post-contrast portable MRI | 6 months
  Blinded neuroradiologists will evaluate the visibility of lesion internal morphology on post-contrast T1-weighted portable MRI images using a standardized 5-point Likert scale (1 = non-visible, 5 = clearly visible). Scores will be summarized using descriptive statistics.
Radiologist-rated degree of contrast enhancement of target lesions on portable MRI | 6 months
  Blinded neuroradiologists will rate the degree of lesion contrast enhancement on post-contrast T1-weighted portable MRI images using a standardized 5-point Likert scale (1 = no enhancement, 5 = marked enhancement). Ratings will be summarized descriptively across subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Neurology, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://hyperfinemri.com/